CLINICAL TRIAL: NCT02453594
Title: A Phase II Clinical Trial of MK-3475 (Pembrolizumab) in Subjects With Relapsed or Refractory (R/R) Classical Hodgkin Lymphoma (cHL)
Brief Title: Study of Pembrolizumab (MK-3475) in Participants With Relapsed or Refractory Classical Hodgkin Lymphoma (MK-3475-087/KEYNOTE-087)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-087; 153005 (Registry Identifier: JAPIC-CTI); 2014-004482-24 (EudraCT Number)
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Hodgkin Lymphoma
Keywords: PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Hodgkin Disease | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants with RRcHL who failed to achieve a response or progressed after auto-SCT and have relapsed after treatment with or failed to respond to BV post auto-SCT received pembrolizumab, 200 mg, intravenously (IV) every 3 weeks (Q3W) on Day 1 of each 21-day cycle for up to 24 months.
  Interventions: Biological: pembrolizumab
- Cohort 2 (Experimental): Participants with RRcHL who were unable to achieve CR or PR to salvage chemotherapy and did not receive auto-SCT, but have relapsed after treatment with or failed to respond to BV received pembrolizumab, 200 mg, IV Q3W on Day 1 of each 21-day cycle for up to 24 months.
  Interventions: Biological: pembrolizumab
- Cohort 3 (Experimental): Participants with RRcHL who failed to achieve a response to or progressed after auto-SCT and have not received BV post auto-SCT received pembrolizumab, 200 mg, IV Q3W on Day 1 of each 21-day cycle for up to 24 months. These participants may or may not have received BV as part of primary treatment or salvage treatment.
  Interventions: Biological: pembrolizumab

INTERVENTIONS:
Biological: pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
This is a study of pembrolizumab (MK-3475) for participants with relapsed/refractory classical Hodgkin Lymphoma (RRcHL) who: 1) have failed to achieve a response or progressed after autologous stem cell transplant (auto-SCT) and have relapsed after treatment with or failed to respond to brentuximab vedotin (BV) post auto-SCT or 2) were unable to achieve a Complete Response (CR) or Partial Response (PR) to salvage chemotherapy and did not receive auto-SCT, but have relapsed after treatment with or failed to respond to BV or 3) have failed to achieve a response to or progressed after auto-SCT and have not received BV post auto-SCT.

The primary study hypothesis is that treatment with single agent pembrolizumab will result in a clinically meaningful overall response rate.

ELIGIBILITY:
Inclusion criteria:

* Relapsed or refractory de novo classical Hodgkin lymphoma
* Participant may have failed to achieve a response to, progressed after, or be ineligible for autologous stem cell transplant (auto-SCT)
* Participant may have failed to achieve a response or progressed after treatment with brentuximab vedotin or may be brentuximab vedotin naïve
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Measurable disease
* Adequate organ function

Exclusion criteria:

* Diagnosis of immunosuppression or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Prior monoclonal antibody within 4 weeks prior to study Day 1 or chemotherapy, targeted small molecular therapy, or radiation therapy within 2 weeks prior to study Day 1
* Prior allogeneic hematopoietic stem cell transplantation
* Known clinically active central nervous system involvement
* Known additional malignancy that is progressing or requires active treatment
* Has a known history of Human Immunodeficiency Virus (HIV)
* Has known active Hepatitis B (HBV) or Hepatitis C (HCV)
* Active autoimmune disease requiring systemic treatment in past 2 years
* Has a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Armand P, Zinzani PL, Lee HJ, Johnson NA, Brice P, Radford J, Ribrag V, Molin D, Vassilakopoulos TP, Tomita A, von Tresckow B, Shipp MA, Herrera AF, Lin J, Kim E, Chakraborty S, Marinello P, Moskowitz CH. Five-year follow-up of KEYNOTE-087: pembrolizumab monotherapy for relapsed/refractory classical Hodgkin lymphoma. Blood. 2023 Sep 7;142(10):878-886. doi: 10.1182/blood.2022019386. PMID 37319435
- [Derived] Armand P, Zinzani PL, Timmerman J, Johnson NA, Lavie D, Thiagarajan K, Topp BG, Pillai P, Herrera AF. Estimating efficacy of favezelimab plus pembrolizumab relative to pembrolizumab in anti-PD-1-refractory Hodgkin lymphoma. Blood Adv. 2025 Oct 14;9(19):4987-4995. doi: 10.1182/bloodadvances.2024014654. PMID 40668662
- [Derived] Chen R, Zinzani PL, Lee HJ, Armand P, Johnson NA, Brice P, Radford J, Ribrag V, Molin D, Vassilakopoulos TP, Tomita A, von Tresckow B, Shipp MA, Lin J, Kim E, Nahar A, Balakumaran A, Moskowitz CH. Pembrolizumab in relapsed or refractory Hodgkin lymphoma: 2-year follow-up of KEYNOTE-087. Blood. 2019 Oct 3;134(14):1144-1153. doi: 10.1182/blood.2019000324. Epub 2019 Aug 13. PMID 31409671
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- [Derived] von Tresckow B, Fanale M, Ardeshna KM, Chen R, Meissner J, Morschhauser F, Moskowitz C, Zinzani PL, Giezek H, Balakumaran A, Vo TT, Raut M, Brice P. Patient-reported outcomes in KEYNOTE-087, a phase 2 study of pembrolizumab in patients with classical Hodgkin lymphoma. Leuk Lymphoma. 2019 Nov;60(11):2705-2711. doi: 10.1080/10428194.2019.1602262. Epub 2019 Apr 23. PMID 31012356
- [Derived] Chen R, Zinzani PL, Fanale MA, Armand P, Johnson NA, Brice P, Radford J, Ribrag V, Molin D, Vassilakopoulos TP, Tomita A, von Tresckow B, Shipp MA, Zhang Y, Ricart AD, Balakumaran A, Moskowitz CH; KEYNOTE-087. Phase II Study of the Efficacy and Safety of Pembrolizumab for Relapsed/Refractory Classic Hodgkin Lymphoma. J Clin Oncol. 2017 Jul 1;35(19):2125-2132. doi: 10.1200/JCO.2016.72.1316. Epub 2017 Apr 25. PMID 28441111
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males and females with relapsed or refractory de novo classical Hodgkin lymphoma (RRcHL) of at least 18 years of age were enrolled in this study.
Groups:
- Cohort 1: Participants with RRcHL who failed to achieve a response or progressed after auto-stem cell transplant (SCT) and have relapsed after treatment with or failed to respond to brentuximab vedotin (BV) post auto-SCT received pembrolizumab, 200 mg, intravenously (IV) every 3 weeks (Q3W) on Day 1 of each 21-day cycle up to 35 cycles, for up to 24 months.
- Cohort 2: Participants with RRcHL who were unable to achieve Complete Response (CR) or Partial Response (PR) to salvage chemotherapy and did not receive auto-SCT, but have relapsed after treatment with or failed to respond to BV received pembrolizumab, 200 mg, IV Q3W on Day 1 of each 21-day cycle up to 35 cycles, for up to 24 months.
- Cohort 3: Participants with RRcHL who failed to achieve a response to or progressed after auto-SCT and have not received BV post auto-SCT received pembrolizumab, 200 mg, IV Q3W on Day 1 of each 21-day cycle, up to 35 cycles for up to 24 months. These participants may or may not have received BV as part of primary treatment or salvage treatment.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started (Randomized) | 69 | 81 | 61
Treated | 69 | 81 | 60
Second Course Pembrolizumab | 10 | 7 | 3
Completed | 0 | 0 | 0
Not Completed | 69 | 81 | 61
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Cohort Was Closed | 17 | 21 | 14
Not completed — Death | 20 | 24 | 16
Not completed — Lost to Follow-up | 6 | 14 | 2
Not completed — Physician Decision | 2 | 4 | 0
Not completed — Site Terminated by Sponsor | 1 | 0 | 1
Not completed — Transitioned to Extension Study | 16 | 9 | 16
Not completed — Withdrawal by Subject | 7 | 9 | 11

BASELINE CHARACTERISTICS:
Population: Treated participants.
Groups:
- Cohort 1: Participants with RRcHL who failed to achieve a response or progressed after auto-SCT and have relapsed after treatment with or failed to respond to BV post auto-SCT received pembrolizumab, 200 mg, intravenously (IV) every 3 weeks (Q3W) on Day 1 of each 21-day cycle up to 35 cycles, for up to 24 months.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 69 | 81 | 60 | 210
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.0 (10.9) | 42.3 (17.4) | 36.8 (13.4) | 39.0 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 38 | 26 | 97
  Male | 36 | 43 | 34 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 3 | 15
  Not Hispanic or Latino | 43 | 63 | 48 | 154
  Unknown or Not Reported | 19 | 13 | 9 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 7 | 4 | 1 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 7
  White | 57 | 73 | 55 | 185
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by BICR Based on IWG Criteria
Description: ORR is the percentage of participants who had a complete response (CR) or partial response (PR) prior to disease progression based on the International Working Group (IWG) criteria using blinded independent central review (BICR). CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. The point estimate and 95% 2-sided exact confidence interval (CI) used the Clopper-Pearson method. An exact binomial test was conducted for each cohort versus a fixed control rate for each cohort. It is hypothesized that ORR will be greater than 20% in each of the 3 cohorts.
Time Frame: Up to approximately 99 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 69 | 81 | 60
Percentage of participants | 78.3 [66.7 to 87.3] | 64.2 [52.8 to 74.6] | 73.3 [60.3 to 83.9]

2. Primary Outcome: Percentage of Participants Experiencing at Least One Adverse Event (AE)
Description: An adverse event (AE) is any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study
Time Frame: Up to 27 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 69 | 81 | 60
Percentage of Participants | 98.6 | 98.8 | 95.0

3. Primary Outcome: Percentage of Participants Discontinuing Study Drug Due to AEs
Description: An AE is any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study
Time Frame: Up to 24 months
Population: All allocated participants who received at least 1 dose of study treatment
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 69 | 81 | 60
Percentage of Participants | 11.6 | 6.2 | 8.3

4. Secondary Outcome: Overall Response Rate (ORR) by BICR Based on Lugano Criteria
Description: ORR is the percentage of participants who had a CR or PR prior to disease progression based on the Lugano criteria using BICR. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. The point estimate and 95% 2-sided exact confidence interval (CI) used the Clopper-Pearson method. An exact binomial test was conducted for each cohort versus a fixed control rate for each cohort.
Time Frame: Up to approximately 99 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 69 | 81 | 60
Percentage of participants | 82.6 [71.6 to 90.7] | 67.9 [56.6 to 77.8] | 68.3 [55.0 to 79.7]

5. Secondary Outcome: Overall Response Rate (ORR) Assessed by Investigator Based on IWG Criteria
Description: ORR is the percentage of participants who had a CR or PR prior to disease progression assessed by the investigator using IWG criteria. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. The point estimate and 95% 2-sided exact confidence interval (CI) used the Clopper-Pearson method. An exact binomial test was conducted for each cohort versus a fixed control rate for each cohort.
Time Frame: Up to approximately 99 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 69 | 81 | 60
Percentage of participants | 72.5 [60.4 to 82.5] | 66.7 [55.3 to 76.8] | 71.7 [58.6 to 82.5]

6. Secondary Outcome: Complete Remission Rate (CRR) by BICR Based on IWG Criteria
Description: CRR is the percentage of participants with complete remission as demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes based on the IWG criteria using BICR. The analysis consisted of the point estimate and 95% 2-sided exact CI, separately by Cohort using the Clopper-Pearson method. Additional analyses were based on site assessment and by central review using the Lugano (2014) criteria.
Time Frame: Up to approximately 99 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 69 | 81 | 60
Percentage of participants | 24.6 | 25.9 | 33.3

7. Secondary Outcome: Complete Remission Rate (CRR) by BICR Based on Lugano Criteria
Description: CRR is the percentage of participants with complete remission as demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes based on the Lugano criteria using BICR. The analysis consisted of the point estimate and 95% 2-sided exact CI, separately by Cohort using the Clopper-Pearson method. Additional analyses were based on site assessment and by central review using the Lugano (2014) criteria.
Time Frame: Up to approximately 99 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 69 | 81 | 60
Percentage of participants | 34.8 | 28.4 | 35.0

8. Secondary Outcome: Complete Remission Rate (CRR) Assessed by Investigator Based on IWG Criteria
Description: CRR is the percentage of participants with complete remission as demonstrated by disappearance of all evidence of disease in the bone marrow, spleen, liver, and lymph nodes assessed by the investigator using IWG criteria. The analysis consisted of the point estimate and 95% 2-sided exact CI, separately by Cohort using the Clopper-Pearson method. Additional analyses were based on site assessment and by central review using the Lugano (2014) criteria.
Time Frame: Up to approximately 99 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 69 | 81 | 60
Percentage of participants | 42.0 | 32.1 | 43.3

9. Secondary Outcome: Progression-free Survival (PFS) Based on BICR
Description: PFS is the time from first dose to the first documented progressive disease (PD) or death due to any cause, whichever occurs first based on BICR. For those who have PD, the true date of disease progression was approximated by the date of the first assessment at which PD is objectively documented per IWG criteria, regardless of discontinuation of study drug. Death is always considered as a confirmed PD event. The non-parametric Kaplan-Meier method was used to estimate the PFS curve with missing data censored at last assessment.
Time Frame: Up to approximately 99 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 69 | 81 | 60
Months | 16.5 [12.0 to 30.3] | 11.1 [7.5 to 13.7] | 19.7 [10.8 to 32.9]

10. Secondary Outcome: Progression-free Survival (PFS) Assessed by the Investigator
Description: PFS is the time from first dose to the first documented progressive disease (PD) or death due to any cause, whichever occurs first assessed by the investigator based on the IWG criteria. For those who have PD, the true date of disease progression was approximated by the date of the first assessment at which PD is objectively documented per IWG criteria, regardless of discontinuation of study drug. Death is always considered as a confirmed PD event. The non-parametric Kaplan-Meier method was used to estimate the PFS curve with missing data censored at last assessment.
Time Frame: Up to approximately 99 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 69 | 81 | 60
Months | 24.9 [13.9 to 33.9] | 13.9 [10.9 to 22.4] | 22.0 [11.1 to 30.3]

11. Secondary Outcome: Duration of Response (DOR) Based on BICR
Description: DOR for the subgroup of participants who achieved a CR or PR by independent central review, is the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of PD or to death due to any cause, whichever comes first based on BICR. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. The analysis used the Kaplan-Meier method, with participants with response censored at their last assessment, and there was no progressive disease at the time of the last disease assessment.
Time Frame: Up to approximately 99 months
Population: All allocated participants who received at least 1 dose of study treatment and had a CR or PR response.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 54 | 52 | 44
Months | 25.0 [0.0 to 88.8] | 11.1 [0.0 to 86.2] | 24.4 [0.0 to 88.3]

12. Secondary Outcome: Duration of Response (DOR) Assessed by the Investigator
Description: DOR for the subgroup of participants who achieved a CR or PR by independent central review, is the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of PD or to death due to any cause, whichever comes first assessed by the investigator based on the IWG criteria. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. The analysis used the Kaplan-Meier method, with participants with response censored at their last assessment, and there was no progressive disease at the time of the last disease assessment.
Time Frame: Up to approximately 99 months
Population: All allocated participants who received at least 1 dose of study treatment and had a CR or PR response.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 50 | 54 | 43
Months | 25.0 [0.0 to 88.8] | 16.4 [0.0 to 86.1] | 24.7 [2.8 to 91.2]

13. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from the first dose to death due to any cause. The Kaplan-Meier method was used to estimate the survival curve, separately by Cohort with missing data censored at last assessment.
Time Frame: Up to approximately 99 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 69 | 81 | 60
Months | NA [NA to NA] — NA means median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA means median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA means median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event.

ADVERSE EVENTS:
Time Frame: Up to approximately 99 months.
Description: The population analyzed for all-cause mortality consisted of all allocated participants. The population for AEs consisted of all allocated participants who received at least 1 dose of study treatment. Per protocol disease progression of cancer was not considered an AE unless related to study drug. Therefore the following AE preferred terms not related to the drug were excluded: Neoplasm progression, Malignant neoplasm progression and Disease progression.
Groups:
- Cohort 1 (First Course): Participants with RRcHL who failed to achieve a response or progressed after auto-stem cell transplant (SCT) and have relapsed after treatment with or failed to respond to brentuximab vedotin (BV) post auto-SCT received pembrolizumab, 200 mg, intravenously (IV) every 3 weeks (Q3W) on Day 1 of each 21-day cycle up to 35 cycles, for up to 24 months.
- Cohort 2 (First Course): Participants with RRcHL who were unable to achieve Complete Response (CR) or Partial Response (PR) to salvage chemotherapy and did not receive auto-SCT, but have relapsed after treatment with or failed to respond to BV received pembrolizumab, 200 mg, IV Q3W on Day 1 of each 21-day cycle up to 35 cycles, for up to 24 months.
- Cohort 3 (First Course): Participants with RRcHL who failed to achieve a response to or progressed after auto-SCT and have not received BV post auto-SCT received pembrolizumab, 200 mg, IV Q3W on Day 1 of each 21-day cycle up to 35 cycles, for up to 24 months. These participants may or may not have received BV as part of primary treatment or salvage treatment.
- Cohort 1 (Second Course): Eligible participants allocated to the pembrolizumab first course in Cohort 1 who stopped (or completed) initial treatment with pembrolizumab after attaining confirmed CR, initiated a second course of pembrolizumab at the investigator's discretion at 200 mg on Day 1 of each 3 week cycle (Q3W) for up to 17 cycles up to approximately an additional year.
- Cohort 2 (Second Course): Eligible participants allocated to the pembrolizumab first course in Cohort 2 who stopped (or completed) initial treatment with pembrolizumab after attaining confirmed CR, initiated a second course of pembrolizumab at the investigator's discretion at 200 mg on Day 1 Q3W for up to 17 cycles up to approximately an additional year.
- Cohort 3 (Second Course): Eligible participants allocated to the pembrolizumab first course in Cohort 3 who stopped (or completed) initial treatment with pembrolizumab after attaining confirmed CR, initiated a second course of pembrolizumab at the investigator's discretion at 200 mg on Day 1 Q3W for up to 17 cycles up to approximately an additional year.
Arm/Group | Cohort 1 (First Course) | Cohort 2 (First Course) | Cohort 3 (First Course) | Cohort 1 (Second Course) | Cohort 2 (Second Course) | Cohort 3 (Second Course)
All-Cause Mortality (participants affected / at risk) | 21/69 | 28/81 | 19/61 | 2/10 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 15/69 | 18/81 | 15/60 | 0/10 | 1/7 | 0/3
Other Adverse Events (participants affected / at risk) | 68/69 | 76/81 | 56/60 | 10/10 | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (First Course) (N=69) | Cohort 2 (First Course) (N=81) | Cohort 3 (First Course) (N=60) | Cohort 1 (Second Course) (N=10) | Cohort 2 (Second Course) (N=7) | Cohort 3 (Second Course) (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (5) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (First Course) (N=69) | Cohort 2 (First Course) (N=81) | Cohort 3 (First Course) (N=60) | Cohort 1 (Second Course) (N=10) | Cohort 2 (Second Course) (N=7) | Cohort 3 (Second Course) (N=3)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 8 (8) | 5 (6) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (6) | 4 (6) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 3 (3) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 8 (9) | 13 (14) | 12 (15) | 0 (0) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Scleral hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 5 (5) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (12) | 11 (11) | 3 (23) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 20 (37) | 12 (19) | 11 (17) | 2 (2) | 4 (7) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 16 (25) | 11 (15) | 11 (32) | 1 (1) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 4 (5) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 16 (22) | 9 (11) | 13 (20) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 6 (8) | 9 (11) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Catheter site erosion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (4) | 2 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 4 (4) | 5 (5) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 15 (16) | 17 (19) | 16 (19) | 3 (3) | 1 (2) | 1 (2)
Influenza like illness (General disorders) | 7 (9) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 27 (48) | 18 (22) | 16 (17) | 4 (5) | 1 (1) | 1 (1)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 6 (6) | 4 (8) | 7 (11) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 12 (15) | 16 (16) | 7 (11) | 2 (3) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 5 (5) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 5 (6) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 8 (8) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 7 (11) | 9 (12) | 5 (9) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 23 (33) | 7 (7) | 12 (22) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (10) | 6 (6) | 5 (7) | 1 (1) | 0 (0) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 6 (6) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (12) | 3 (3) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (12) | 3 (3) | 1 (1) | 1 (4) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 5 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 4 (6) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (5) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 3 (3) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 6 (6) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (4) | 1 (2) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (5) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (20) | 12 (14) | 6 (10) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (11) | 12 (13) | 5 (6) | 3 (3) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (12) | 1 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 5 (7) | 5 (8) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Tumour inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (19) | 6 (11) | 10 (11) | 2 (2) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (4) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 6 (8) | 7 (7) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (26) | 22 (37) | 14 (19) | 2 (3) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (19) | 10 (16) | 7 (13) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 8 (8) | 8 (14) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 7 (8) | 9 (11) | 1 (1) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 1 (1) | 4 (6) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tonsillar exudate (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (16) | 11 (18) | 7 (8) | 3 (3) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 12 (15) | 9 (11) | 10 (14) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT02453594/Prot_SAP_000.pdf